CLINICAL TRIAL: NCT04617860
Title: A Multicenter, Open-label Extension Study to Evaluate the Safety, Pharmacodynamics, and Clinical Effects of WVE-120102 in Patients With Huntington's Disease
Brief Title: Open-label Extension Study to Evaluate the Safety and Tolerability of WVE-120102 in Patients With Huntington's Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVE-HDSNP2-002
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- WVE-120102 (Dose A) (Experimental)
  Interventions: Drug: WVE-120102

INTERVENTIONS:
Drug: WVE-120102 — WVE-120102 is a stereopure antisense oligonucleotide. It is administered monthly via intrathecal injection.

SUMMARY:
WVE-HDSNP2-002 is an open-label extension (OLE) study to evaluate the safety, tolerability, PK, PD, and clinical effects of WVE-120102 in adult patients with early manifest HD who carry a targeted single nucleotide polymorphism, rs362331 (SNP2). To participate in the study, patients must have completed the Phase 1b/2a clinical study WVE-HDSNP2-001.

ELIGIBILITY:
Inclusion Criteria:

1. Patient successfully completed the Phase 1b/2a study with WVE-120102, WVE-HDSNP2-001.

Exclusion Criteria:

1. Received an investigational drug other than WVE-120102, including an investigational oligonucleotide, within the past 1 year or 5 half-lives of the drug, whichever is longer.
2. Inability to undergo brain MRI (with or without sedation).
3. Clinically significant medical finding on the physical examination other than HD that, in the judgment of the Investigator, will make the patient unsuitable for participation in and/or completion of the study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — WAVE Life Sciences
Locations (20):
- Australia (7):
  - Westmead Hospital, Sydney, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Royal Melbourne Hospital, Carlton, Victoria
  - Monash Health, Clayton, Victoria
  - Alfred Health, Melbourne, Victoria
  - Calvary Health Care Bethlehem, Parkdale, Victoria
  - North Metropolitan Health Service, Perth, Western Australia
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - Centre For Movement Disorders, Toronto, Ontario
  - Centre Hospitalier de l-Universite de Montreal, Montreal, Quebec
- Denmark (3):
  - Aarhus Universitets Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital and University of Southern Denmark, Odense
- France (2):
  - Hospital Henri Mondor, Créteil
  - Institut du Cerveau et de la Moelle Epinière, Paris
- George-Huntington-Institut GmbH, Münster, Germany
- Poland (2):
  - Szpital Sw. Wojciecha, Gdansk
  - Instytut Psychiatrii i Neurologii, Warsaw
- United Kingdom (2):
  - Royal Devon and Exeter Hospital NHS Trust, Exeter, Devon
  - Queen Elizabeth University Hospital - PPDS, Glasgow, Glasgow City

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the original OLE study protocol, patients who were in the 2 and 4 mg dose cohorts in the Phase 1b/2a study were to be enrolled into the 4 or 8 mg dose group in this study. Patients in the 8 and 16 mg dose cohorts in WVE-HDSNP1-001 continued to receive that dose. As of Amendment 2.0 of this protocol, all new patients were to be enrolled at a dose level of at least 16 mg. All current patents were dose modified to 16 or 32 mg.
Groups:
- 4 mg WVE-120102: Enrolled at 4 mg WVE-120102 dose level
- 8 mg WVE-120102: Enrolled at 8 mg WVE-120102 dose level
- 16 mg WVE-120102: Enrolled at 16 mg WVE-120102 dose level
Period: Overall Study
Arm/Group | 4 mg WVE-120102 | 8 mg WVE-120102 | 16 mg WVE-120102
Started | 8 | 10 | 18
Dose Modified to 8 mg | 8 | 1 | 0
Dose Modified to 16 mg | 8 | 9 | 8
Dose Modified to 32 mg | 2 | 4 | 11
Completed | 0 | 0 | 0
Not Completed | 8 | 10 | 18
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Sponsor Decision | 0 | 3 | 1
Not completed — Termination of Study by Sponsor | 8 | 4 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 mg WVE-120102 | 8 mg WVE-120102 | 16 mg WVE-120102 | Total
Number analyzed (Participants) | 8 | 10 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 16 | 33
  >=65 years | 1 | 0 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 7 | 16
  Male | 5 | 4 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 10 | 18 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 10 | 18 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 1 | 12 | 21
  Denmark | 0 | 5 | 0 | 5
  Poland | 0 | 4 | 5 | 9
  Australia | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Patients With Treatment-emergent Adverse Events (TEAEs)
Time Frame: Day 1 to Study Termination (maximum of 12 monthly doses)
Population: Patients treated at more than one dose level (e.g., initial dose and after dose modification) are included in each applicable dose group. Adverse events are counted in the dose the patient was receiving at the time of onset.
Measure: Count of Participants; unit: Participants
Groups:
- 4 mg WVE-120102: Received 4 mg WVE-120102 at any point in the study
- 8 mg WVE-120102: Received 8 mg WVE-120102 at any point in the study
- 16 mg WVE-120102: Received 16 mg WVE-120102 at any point in the study
- 32 mg WVE-120102: Received 32 mg WVE-120102 at any point in the study
Arm/Group | 4 mg WVE-120102 | 8 mg WVE-120102 | 16 mg WVE-120102 | 32 mg WVE-120102
Number analyzed (Participants) | 8 | 18 | 35 | 17
Participants | 7 | 14 | 34 | 17

2. Primary Outcome: Safety: Number of Patients With a Severe TEAE
Time Frame: Day 1 to Study Termination (maximum of 12 monthly doses)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg WVE-120102 | 8 mg WVE-120102 | 16 mg WVE-120102 | 32 mg WVE-120102
Number analyzed (Participants) | 8 | 18 | 35 | 17
Participants | 0 | 0 | 2 | 5

3. Primary Outcome: Safety: Number of Patients With Serious TEAEs
Time Frame: Day 1 to Study Termination (maximum of 12 monthly doses)
Population: Patients treated at more than one dose level (e.g. initial dose and after dose modification) are included in each applicable dose group. Adverse events are counted in the dose the patient was receiving at the time of onset.
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg WVE-120102 | 8 mg WVE-120102 | 16 mg WVE-120102 | 32 mg WVE-120102
Number analyzed (Participants) | 8 | 18 | 35 | 17
Participants | 0 | 1 | 5 | 3

4. Primary Outcome: Safety and Tolerability: Number of Patients Who Withdraw Due to TEAEs
Time Frame: Day 1 to Study Termination (maximum of 12 monthly doses)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg WVE-120102 | 8 mg WVE-120102 | 16 mg WVE-120102 | 32 mg WVE-120102
Number analyzed (Participants) | 8 | 18 | 35 | 17
Participants | 0 | 1 | 3 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Study Termination (maximum of 12 monthly doses)
Arm/Group | 4 mg WVE-120102 | 8 mg WVE-120102 | 16 mg WVE-120102 | 32 mg WVE-120102
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/18 | 0/35 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/18 | 5/35 | 3/17
Other Adverse Events (participants affected / at risk) | 7/8 | 14/18 | 34/35 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 mg WVE-120102 (N=8) | 8 mg WVE-120102 (N=18) | 16 mg WVE-120102 (N=35) | 32 mg WVE-120102 (N=17)
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Meningitis (Infections and infestations) | 0 | 1 | 1 | 0
Meningitis asceptic (Infections and infestations) | 0 | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 2
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 4 mg WVE-120102 (N=8) | 8 mg WVE-120102 (N=18) | 16 mg WVE-120102 (N=35) | 32 mg WVE-120102 (N=17)
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Paresthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 6 | 2
Fatigue (General disorders) | 0 | 0 | 6 | 4
Pain (General disorders) | 1 | 0 | 3 | 1
Gait disturbance (General disorders) | 0 | 0 | 2 | 1
Injection site erythema (General disorders) | 1 | 0 | 0 | 0
Injection site hypersensitivity (General disorders) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 5 | 2
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 4 | 2
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
CSF protein increased (Investigations) | 0 | 3 | 7 | 4
CSF lymphocyte count increased (Investigations) | 0 | 2 | 5 | 0
CSF test abnormal (Investigations) | 0 | 0 | 0 | 3
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 1
CSF white blood cell count (Investigations) | 0 | 0 | 2 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 2 | 0
Complement factor increased (Investigations) | 0 | 0 | 0 | 1
Dermatologic examination abnormal (Investigations) | 0 | 0 | 0 | 1
Neurological examination abnormal (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 6 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 2 | 6 | 14 | 6
Dizziness (Nervous system disorders) | 0 | 0 | 4 | 3
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 3
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 2
Dyskinesia (Nervous system disorders) | 1 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 2 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 3 | 5
Apathy (Psychiatric disorders) | 0 | 1 | 1 | 0
Behavior disorder (Psychiatric disorders) | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 2 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 2 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 1
Persecutory delusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dysnpoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT04617860/Prot_SAP_000.pdf